CLINICAL TRIAL: NCT03769324
Title: Validation of Osmolarity System: Clinical Usability Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: I-MED Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: IPCT201810
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal Eye Group: Normal eye receiving Osmolarity Test
  Interventions: Diagnostic Test: Osmolarity Test
- DED Group: Dry Eye Disease receiving Osmolarity Test
  Interventions: Diagnostic Test: Osmolarity Test

INTERVENTIONS:
Diagnostic Test: Osmolarity Test — Osmolarity Test

SUMMARY:
Confirmatory trial to validate usability of a new portable osmolarity testing device.

DETAILED DESCRIPTION:
Confirmatory trial at 3 sites in Canada to validate usability of an ocular osmolarity testing device.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent

Exclusion Criteria:

* Ocular pathology (other than Dry Eye)

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dry Eye Disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Osmolarity Level | Baseline
  Osmolarity Level

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Hofmann, PhD, Study Chair — I-MED Pharma, Inc.

IPD SHARING:
Plan to Share IPD: No